CLINICAL TRIAL: NCT02214771
Title: Description of the Use of fidAxomicin in Hospitalized Patients With Documented Clostridium diFficile iNfection and of the managEment of These Patients (DAFNE Study)
Brief Title: Description of the Use of fidAxomicin in Hospitalized Patients With Documented Clostridium diFficile iNfection and of the managEment of These Patients
Acronym: DAFNE
Status: Completed | Type: Observational
Sponsor: Astellas Pharma S.A.S. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: FR-FID-NI-001
Record Dates: First submitted 2014-05-13; First posted 2014-08-12 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile infection CDI; Observational; Fidaxomicin recurrence; France
MeSH Terms: conditions — Clostridium Infections | interventions — Fidaxomicin; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: CDI in patients treated with fidaxomicin: Diagnosed with a CDI and treated with fidaxomicin
  Interventions: Drug: Fidaxomicin
- 2: CDI in patients receiving treatment other than fidaxomicin: Diagnosed with a CDI, regardless of the prescribed treatment (not fidaxomicin)
  Interventions: Drug: Treatment for CDI other than fidaxomicin Type

INTERVENTIONS:
Drug: Fidaxomicin — oral
  Other Names: Dificid; ASP2819; Dificlir
  Groups: 1: CDI in patients treated with fidaxomicin
Drug: Treatment for CDI other than fidaxomicin Type — Oral
  Groups: 2: CDI in patients receiving treatment other than fidaxomicin

SUMMARY:
The study aims to describe the characteristics and the methods of management and follow-up of patients treated with fidaxomicin for Clostridium difficile infection (CDI).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Patient diagnosed with CDI

Exclusion Criteria:

* Patient already included in this study
* Patient is taking part in a clinical trial in the field of CDI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients diagnosed with clostridium difficile infection
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Characteristics of patients treated with fidaxomicin, including demographic data, description of comorbidities and treatment by antibiotherapy | Day 1
Characteristics of the CDI treated with fidaxomicin, including date of CDI diagnosis, department requesting the diagnosis of CDI, methods used, severity of CDI and origin of the case | Day 1

SECONDARY OUTCOMES:
Therapeutic management of the CDI, including the starting date of the treatment, CDI treatment first line and associated treatment | Day 1
  For patients treated with fidaxomicin
Number and timing of recurrences in patients treated with fidaxomicin over a 3-month follow-up period | End of the follow-up (3 months)
Adverse events and serious adverse events occurring on fidaxomicin | End of the follow-up (3 months)
Characteristics of patients diagnosed with CDI, including demographic data and treatment by antibiotherapy | Day 1
  For all patients diagnosed with CDI regardless of treatment
Characteristics of the CDI, including date of CDI diagnosis, Department requesting the diagnosis of CDI, methods used, severity of CDI and origin of the case | Day 1
  For all patients diagnosed with CDI regardless of treatment
Treatment of the CDI including treatment selected and dosage | Day 1
  For all patients diagnosed with CDI regardless of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Scientific Affairs manager, Study Director — Astellas Pharma S.A.S.
Locations (24):
- France (24):
  - Site, Béthune
  - Site, Bordeaux
  - Site, Boulogne-Billancourt
  - Site, Caen
  - Site, Chambéry
  - Site, Clermond-Ferrand
  - Site, Clichy
  - Site, Dijon
  - Site, Garches
  - Site, La Tronche
  - Site, Lille
  - Site, Lyon
  - Site, Marseille
  - Site, Morlaix
  - Site, Mulhouse
  - Site, Nantes
  - Site, Nîmes
  - Site, Orléans
  - Site, Paris
  - Site, Poitiers
  - Site, Reims
  - Site, Rennes
  - Site, Roubaix
  - Site, Soissons

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guery B, Berger P, Gauzit R, Gourdon M, Barbut F; DAFNE study group; Dafne Study Group, Bemer P, Bessede E, Camou F, Cattoir V, Couzigou C, Descamps D, Dinh A, Laurans C, Lavigne JP, Lechiche C, Leflon-Guibout V, Le Monnier A, Levast M, Mootien JY, N'Guyen Y, Piroth L, Prazuck T, Rogeaux O, Roux AL, Vachee A, Vernet Garnier V, Wallet F. A prospective, observational study of fidaxomicin use for Clostridioides difficile infection in France. J Int Med Res. 2021 Jun;49(6):3000605211021278. doi: 10.1177/03000605211021278. PMID 34162264